CLINICAL TRIAL: NCT02549534
Title: Early Detection of Taxane-Induced Neuropathy in Women With Breast Cancer
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Midwest Nursing Research Society (MNRS) (Unknown); Council for the Advancement of Nursing Science (CANS) (Unknown); Indiana Center for Vascular Biology & Medicine (ICVBM) (Unknown); Indiana University School of Medicine (Other)
Responsible Party: Principal Investigator, Victoria L. Champion, Distinguished Professor of Nursing; Edward and Sarah Stam Cullipher Endowed Chair; Associate Director of Cancer Control and Population Sciences, Indiana University Simon Cancer Center (IUSCC), Indiana University
Other Study IDs: 1502603664; F31NR01521201A1 (Other Grant/Funding Number: National Institute of Nursing Research (NIH))
Record Dates: First submitted 2015-09-09; First posted 2015-09-15 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Peripheral Neuropathy
Keywords: Taxane; Neuropathy; Chemotherapy-Induced Peripheral Neuropathy (CIPN); Breast Cancer; Local skin heating; Axon reflex; Axon flare; Total Neuropathy Score (TNS); Laser Doppler Flowmetry (LDF); Laser Speckle Contrast Imaging (LSCI); Full-field laser perfusion imaging (FLPI); Paclitaxel; Taxol
MeSH Terms: conditions — Peripheral Nervous System Diseases; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Women with Breast Cancer (WBC): Defined as women who:
  * Are 18 to 85 years old at the time of enrollment;
  * Have histologically-confirmed, first-time, non-metastatic breast cancer (Stage I-IIIB);
  * Have no history of neurotoxic chemotherapy or radiation treatment at the time of enrollment;
  * Will be receiving weekly paclitaxel (Taxol® or generic paclitaxel), 80-100mg/m2, or bi-weekly (i.e., dose-dense) Taxol, 175 mg/m2, as a part of their treatment regimen OR
  * Will be receiving an anthracycline and cyclophosphamide (AC) therapy followed by weekly or bi-weekly (i.e., dose-dense; 175 mg/m2) paclitaxel (Taxol® or generic paclitaxel, 80-100mg/m2);
  * Are willing to participate in up to four study sessions.
  Interventions: Procedure: Axon Reflexes; Procedure: Axon Flares; Procedure: Self-Reported Signs & Symptoms of CIPN
- Healthy Female Controls (HCs): Defined as women who:
  * Are 18 to 85 years old at the time of study enrollment;
  * Can read, write, and understand English,
  * Are willing to participate in three planned study sessions.
  Interventions: Procedure: Axon Reflexes; Procedure: Axon Flares; Procedure: Self-Reported Signs & Symptoms of CIPN

INTERVENTIONS:
Procedure: Axon Reflexes — *Axon reflexes will be evoked in the palmar surface of the right great toe using local skin heating with a 0.33 cm2 heat probe using the following protocol:
  * Baseline: Heating the skin of the toe for a minimum of 5 minutes at 33*C.
  * Heat Ramp: Increasing the heat in the heat probe to 42*C at approx. 0.1*C/10 sec.
  * Skin Heating: Heating the skin of the toe for 30 minutes 42*C.
  * Heat Ramp: Increasing the heat in the heat probe to 44*C at 0.1*C/10 sec..
  * Skin Heating: Heating the skin for an additional 5 minutes at 44*C.
  The size of the axon reflex during this skin heating protocol will be imaged using Laser Doppler Flowmetry (LDF). In the case that participants develop CIPN on their left side only, the left toe will be substituted.
Procedure: Axon Flares — Axon flares will be generated on the palmar surface of the right great toe using the same local skin heating protocol described above, and imaged using a laser speckle contrast imager (LSCI) (also known as full-field laser perfusion imager, or FLPI).
  Other Names: LDIflare, Heat-Evoked Axon Flare
Procedure: Self-Reported Signs & Symptoms of CIPN — Self-reported signs & symptoms of CIPN such as the presence and location of (1) tingling, (2) numbness, and (3) neuropathic pain, along with information about (4) deficits in vibration thresholds, and (5) loss of deep tendon reflexes will be assessed at each study visit using the 5-item, modified Total Neuropathy Score (mTNS).

SUMMARY:
Purpose: The purpose of the study is to test a new way of measuring nerve damage in women with breast cancer receiving chemotherapy drug paclitaxel (Taxol).

DETAILED DESCRIPTION:
Purpose: The study has four aims;

* The primary aim of the study is to determine whether women who are receiving either weekly Taxol (80-100 mg/m2) or bi-weekly Taxol (i.e.,dose-dense; 175 mg/m2) show deficits in axon-reflex mediated vasodilation (AMV) over the course of six weeks of Taxol therapy similar to those that have been reported in patients with diabetic and genetically-inherited neuropathies.
* The second aim of the study is to determine whether women who are receiving either weekly or dose-dense Taxol develop changes in AMV before developing signs & symptoms of chemotherapy-induced peripheral neuropathy (CIPN) in a way that supports using changes in AMV as an early detection method for small-fiber CIPN.
* A third (exploratory) aim of the study is to determine whether any changes in AMV detected during the study are significantly correlated with self-reported CIPN in a way that would support using changes in AMV as a confirmatory marker for CIPN.
* A final (exploratory) aim of the study is to describe the size of axon reflexes and axon flares in women receiving weekly Taxol before they start their pre-Taxol anthracycline & cyclophosphamide (AC) therapy.

ELIGIBILITY:
Inclusion Criteria for Women with Breast Cancer:

* Age 18-85
* Able to read, write, and understand English
* Diagnosed with histologically-confirmed, first-time, non-metastatic breast cancer (stage I-IIIB)
* No prior exposure to neurotoxic chemotherapy or radiation at the time of enrollment,
* Will be receiving weekly paclitaxel (Taxol® or generic paclitaxel, 80- 100mg/m2) or bi-weekly Taxol (i.e., dose-dense; 175 mg/m2) as a part of their cancer treatment regimen OR
* Will be receiving an anthracycline and cyclophosphamide (AC) followed by weekly paclitaxel (Taxol® or generic paclitaxel, 80-100mg/m2) or bi-weekly Taxol (i.e., dose-dense; 175 mg/m2) as a part of their cancer treatment regimen;

Inclusion Criteria for Healthy Controls:

* Aged 18-85
* Can read, write, and understand English

Exclusion Criteria:

* A history of cardiovascular disease, hypertension, or peripheral arterial/vascular disease;
* Current use of (1) medications/supplements to control blood pressure (e.g. beta-blockers, nitrates, calcium channel blockers, Phosphodiesterase-5 (PGE5) inhibitors) or (2) the use of statins for cholesterol;
* Suspected or diagnosed diabetes (with the exception of gestational diabetes);
* Pre-existing neuropathy, neuropathic pain, or nerve injury;
* Pain or significant arthritis in the toes of either foot;
* Current skin disease or fungal infection of the feet;
* Significant damage or deformity to the feet that would alter blood flow or make it impossible to measure/interpret findings;
* Diagnosed or suspected vasospastic disease such as Raynaud's syndrome;
* Current use of tobacco/tobacco-containing products;
* Diagnosis of restless leg syndrome or other movement disorders that would prevent accurate data from being able to be collected.

In-Study Restrictions:

* No caffeine- or alcohol-containing products for 12 hours prior to their study visit;
* No food for at least one hour prior to blood flow monitoring;
* No non-steroidal anti-inflammatory drugs (NSAIDS) for 24 hours prior to study visits unless directed by a physician to do so.

(Note: These restrictions are designed to improve the rigor and quality of the data, but non-compliance will not be grounds for study exclusion; adherence to these restrictions will be monitored during self-report).

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult women with breast cancer (WBC) and healthy female controls (HCs)
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2015-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Differences in the mean size of axon reflexes between healthy women and women with breast cancer BEFORE starting Taxol. | Day 1 (before participant's 1st Taxol infusion).
  * Hypothesis: (Cross-Sectional): There WILL NOT be a significant difference in the mean size of axon reflexes (expressed as a %CVCmax) in the great toe between healthy women and women with breast cancer before they start Taxol (i.e., Day 1).
  * Definitions/Notes: The mean size of axon reflexes will be determined by averaging the peak laser doppler values (in tissue perfusion units (TPUs)) that occur during a stable 30-90 second period after increasing the probe temperature to 42*C. The maximum circulatory vascular conductance (%CVCmax) for each participant will be determined by dividing the raw TPU values by the participant's mean arterial blood pressure (MAP) during the axon reflex. The size of axon reflexes for each group will be then calculated by averaging the %CVCmax values corresponding to each individual's axon reflex for each group at that time point. Differences between groups in the size of axon reflexes at Day 1 will be compared using two-tailed t-tests, α=0.05.
Differences in the mean size of axon reflexes between healthy women and women with breast cancer DURING Taxol therapy. | Day 14 (week two of Taxol therapy) and Day 42 (week six of Taxol therapy).
  * Hypothesis (Cross-Sectional): There WILL be a significant difference in the mean size of axon reflexes generated on the palmar surface of the right great toe between healthy controls and women with breast cancer during their initial six weeks of Taxol therapy (i.e., day 14 and 42, respectively).
  * Notes: The mean size of axon reflexes during Taxol therapy will be determined by averaging the size of axon reflexes for participants in each group at day 14 and 42, respectively. Differences between groups in the size of axon reflexes at day 14 and 42 will be compared using two-tailed t-tests, α=0.05.
Differences in the mean size of axon reflexes OVER TIME for women with breast during the initial six weeks of Taxol therapy. | Day 1 (before participant's 1st Taxol infusion), day 14 (week two of Taxol therapy) and day 42 (week six of Taxol therapy).
  * Hypothesis (Longitudinal): There WILL be a significant difference in the mean size of axon reflexes generated on the palmar surface of the great toe of women with breast cancer from (a) day 1 to day 14, (b) day 14 to day 42, and from (c) day 1 to day 42.
  * Note: Differences in mean size of axon reflexes over the course of Taxol therapy will be calculated using repeated-measures analysis of covariance (RM-ANCOVA).
Differences in the mean size of axon reflexes between healthy female controls OVER TIME the six-week study period. | Day 1 (before participant's 1st Taxol infusion), Day 14 (week two of Taxol therapy) and Day 42 (week six of Taxol therapy).
  * Hypothesis (Longitudinal): There WILL NOT be a significant difference in the size of axon reflexes on the palmar surface of the great toe of healthy female controls from(a) day 1 to day 14, (b) day 14 to day 42, and from (c) day 1 to day 42.
  * Note: Differences in mean size of axon reflexes over the course of Taxol therapy will be calculated using repeated-measures analysis of covariance (RM-ANCOVA).

SECONDARY OUTCOMES:
Differences in the mean size of heat-evoked axon flares between healthy women and women with breast cancer BEFORE starting Taxol therapy. | Day 1 (before participant's 1st Taxol infusion).
  * Hypothesis (Cross-Sectional): There WILL NOT be a significant difference in the mean size of heat-evoked axon flares generated on the palmar surface of the great toe between healthy women and women with breast cancer before starting Taxol therapy (day 1).
  * Note: A "heat-evoked axon flare" is defined as the area of increased cutaneous blood flow surrounding heat probe that is at least three standard deviations (3SD) above blood flow measured during prior to local skin heating. The size of each axon flare will be expressed in centimeters squared (cm2). The mean size of axon flares for each group will be calculated by averaging the size of axon flares for healthy women at baseline and the size of axon flares for women with breast cancer at day 1 (before starting Taxol). Differences in the mean size of axon flares between both groups at day 1 will be compared using two-tailed t-tests, α=0.05.
Differences in the mean size of heat-evoked axon flares between healthy women and women with breast cancer DURING six weeks of study visits. | Day 14 (week two of Taxol therapy) and Day 42 (week six of Taxol therapy).
  * Hypothesis (Cross-Sectional): There WILL be a significant difference in the mean size of heat-evoked axon flares generated on the palmar surface of the great toe between healthy controls and women with breast cancer DURING Taxol therapy at day 14 and 42 (respectively).
  * Note: Differences in the size of heat-evoked axon flares between healthy women and women with breast cancer at days 14 and 42 (respectively) will be compared using separate, two-tailed t-tests, α=0.05.
Differences in the mean size of heat-evoked axon flares between women with breast cancer DURING their initial six weeks of Taxol therapy. | Day 1 (before participant's 1st Taxol infusion), Day 14 (week two of Taxol therapy) and Day 42 (week six of Taxol therapy).
  * Hypothesis (Longitudinal): There WILL be a significant difference in the mean size of heat-evoked axon flares generated on the palmar surface of great toe of women with breast cancer receiving Taxol from (a) day 1 to day 14, (b) day 14 to day 42, and from (c) day 1 to day 42.
  * Differences in the size of heat-evoked axon flares during Taxol therapy will be evaluated using repeated-measures analysis of variance (RM-ANOVA).
Differences in the size of heat-evoked axon flares for healthy women during the six-week study period. | Day 1 (before participant's 1st Taxol infusion), Day 14 (week two of Taxol therapy) and Day 42 (week six of Taxol therapy).
  * Hypothesis (Longitudinal): There WILL NOT be a significant difference in the size of heat-evoked axon flares (in cm2) generated on the great toe of healthy women from (a) day 1 to day 14, (b) day 14 to day 42, and from (c) day 1 to day 42.
  * Differences in the size of heat-evoked axon flares during Taxol therapy will be evaluated using RM-ANOVA.

OTHER OUTCOMES:
Correlations between the size of axon reflexes (expressed in %CVCmax) and the average modified-Total Neuropathy (m-TNS) score for women with breast cancer AT EACH TIMEPOINT during Taxol Therapy. | Day 1 (before participant's 1st Taxol infusion), Day 14 (week two of Taxol therapy) and Day 42 (week six of Taxol therapy).
  * Hypothesis: There WILL BE a statistically significant, inverse correlation between (a) the size of axon reflexes generated on the great toe and (b) the mean total m-TNS scores for women with breast cancer receiving Taxol at Days 1, 14, and 42 (respectively).
  * Note: The 'size of axon reflexes' will be defined using the criteria above. The 'average m-TNS score' will be calculated by averaging the total Modified-Total Neuropathy Score (m-TNS) score (1-20) for each woman with breast cancer, at each time point. Pearson R will be used to determine the magnitude, direction, and statistical significance of bivariate correlations between (a) axon reflex size and (b) average mTNS scores for women with breast cancer receiving Taxol at each study time point.
Correlation between the size of axon reflexes (expressed in %CVCmax) and the average modified Total Neuropathy Score (TNS) for healthy women AT EACH TIMEPOINT during the six-week study period. | Day 1 (before participant's 1st Taxol infusion), Day 14 (week two of Taxol therapy) and Day 42 (week six of Taxol therapy).
  * Hypothesis (Cross-Sectional): There WILL NOT be a significant inverse correlation between the size of axon reflexes generated on the palmar surface of the great toe and healthy women's mean total m-TNS scores at Days 1, 14, and 42 (respectively). (Note: Definitions and analyses are the same as above.)
Correlation between (a) the size of heat-evoked axon flares (in cm2) and (b) the average modified-Total Neuropathy Score (mTNS) for women with breast cancer AT EACH TIMEPOINT during Taxol Therapy. | Day 1 (before participant's 1st Taxol infusion), Day 14 (week two of Taxol therapy) and Day 42 (week six of Taxol therapy).
  * Hypothesis: There WILL be a statistically significant, inverse correlation between (a) the size of heat-evoked axon flares generated on the palmar surface of the great toe and (b) mean total mTNS scores for women with breast cancer receiving weekly Taxol at Days 1, 14, and 42 (respectively).(Note: Definitions and analyses are the same as above.)
Correlation between (a) the size of heat-evoked axon flares (in cm2) and (b) the average modified-Total Neuropathy Score (mTNS) for healthy women AT EACH TIMEPOINT during Taxol Therapy. | Day 1 (before participant's 1st Taxol infusion), Day 14 (week two of Taxol therapy) and Day 42 (week six of Taxol therapy).
  * Hypothesis: There WILL NOT be a statistically significant, inverse correlation between (a) the size of heat-evoked axon flares generated on the palmar surface of the great toe and (2) healthy women's mean total m-TNS scores at Days 1, 14, and 42 (respectively). (Note: Definitions and analyses are the same as above.)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria L. Champion, PhD,RN,FAAN, Principal Investigator — Indiana University School of Medicine
Locations (2):
- United States (2):
  - Indiana University Melvin and Bren Simon Cancer Center (IUSCC), Indianapolis, Indiana
  - Syndney & Lois Eskenazi Health Center, Indianapolis, Indiana

REFERENCES:
- [Background] Golan-Vered Y, Pud D. Chemotherapy-induced neuropathic pain and its relation to cluster symptoms in breast cancer patients treated with paclitaxel. Pain Pract. 2013 Jan;13(1):46-52. doi: 10.1111/j.1533-2500.2012.00554.x. Epub 2012 Apr 26. PMID 22533683
- [Background] Hershman DL, Weimer LH, Wang A, Kranwinkel G, Brafman L, Fuentes D, Awad D, Crew KD. Association between patient reported outcomes and quantitative sensory tests for measuring long-term neurotoxicity in breast cancer survivors treated with adjuvant paclitaxel chemotherapy. Breast Cancer Res Treat. 2011 Feb;125(3):767-74. doi: 10.1007/s10549-010-1278-0. Epub 2010 Dec 3. PMID 21128110
- [Background] Wolf SL, Barton DL, Qin R, Wos EJ, Sloan JA, Liu H, Aaronson NK, Satele DV, Mattar BI, Green NB, Loprinzi CL. The relationship between numbness, tingling, and shooting/burning pain in patients with chemotherapy-induced peripheral neuropathy (CIPN) as measured by the EORTC QLQ-CIPN20 instrument, N06CA. Support Care Cancer. 2012 Mar;20(3):625-32. doi: 10.1007/s00520-011-1141-9. Epub 2011 Apr 12. PMID 21479990
- [Background] Forsyth PA, Balmaceda C, Peterson K, Seidman AD, Brasher P, DeAngelis LM. Prospective study of paclitaxel-induced peripheral neuropathy with quantitative sensory testing. J Neurooncol. 1997 Oct;35(1):47-53. doi: 10.1023/a:1005805907311. PMID 9266440
- [Background] O'Shaughnessy J, Gradishar WJ, Bhar P, Iglesias J. Nab-paclitaxel for first-line treatment of patients with metastatic breast cancer and poor prognostic factors: a retrospective analysis. Breast Cancer Res Treat. 2013 Apr;138(3):829-37. doi: 10.1007/s10549-013-2447-8. Epub 2013 Apr 6. PMID 23563958
- [Background] Park SB, Goldstein D, Krishnan AV, Lin CS, Friedlander ML, Cassidy J, Koltzenburg M, Kiernan MC. Chemotherapy-induced peripheral neurotoxicity: a critical analysis. CA Cancer J Clin. 2013 Nov-Dec;63(6):419-37. doi: 10.3322/caac.21204. PMID 24590861
- [Background] Osmani K, Vignes S, Aissi M, Wade F, Milani P, Levy BI, Kubis N. Taxane-induced peripheral neuropathy has good long-term prognosis: a 1- to 13-year evaluation. J Neurol. 2012 Sep;259(9):1936-43. doi: 10.1007/s00415-012-6442-5. Epub 2012 Feb 17. PMID 22349867
- [Background] Pignata S, De Placido S, Biamonte R, Scambia G, Di Vagno G, Colucci G, Febbraro A, Marinaccio M, Lombardi AV, Manzione L, Carteni G, Nardi M, Danese S, Valerio MR, de Matteis A, Massidda B, Gasparini G, Di Maio M, Pisano C, Perrone F. Residual neurotoxicity in ovarian cancer patients in clinical remission after first-line chemotherapy with carboplatin and paclitaxel: the Multicenter Italian Trial in Ovarian cancer (MITO-4) retrospective study. BMC Cancer. 2006 Jan 7;6:5. doi: 10.1186/1471-2407-6-5. PMID 16398939
- [Background] Speck RM, Sammel MD, Farrar JT, Hennessy S, Mao JJ, Stineman MG, DeMichele A. Impact of chemotherapy-induced peripheral neuropathy on treatment delivery in nonmetastatic breast cancer. J Oncol Pract. 2013 Sep;9(5):e234-40. doi: 10.1200/JOP.2012.000863. Epub 2013 Apr 30. PMID 23943894
- [Background] Boddy AV, Plummer ER, Todd R, Sludden J, Griffin M, Robson L, Cassidy J, Bissett D, Bernareggi A, Verrill MW, Calvert AH. A phase I and pharmacokinetic study of paclitaxel poliglumex (XYOTAX), investigating both 3-weekly and 2-weekly schedules. Clin Cancer Res. 2005 Nov 1;11(21):7834-40. doi: 10.1158/1078-0432.CCR-05-0803. PMID 16278406
- [Background] Sarosy G, Kohn E, Stone DA, Rothenberg M, Jacob J, Adamo DO, Ognibene FP, Cunnion RE, Reed E. Phase I study of taxol and granulocyte colony-stimulating factor in patients with refractory ovarian cancer. J Clin Oncol. 1992 Jul;10(7):1165-70. doi: 10.1200/JCO.1992.10.7.1165. PMID 1376773
- [Background] Rowinsky EK, Chaudhry V, Forastiere AA, Sartorius SE, Ettinger DS, Grochow LB, Lubejko BG, Cornblath DR, Donehower RC. Phase I and pharmacologic study of paclitaxel and cisplatin with granulocyte colony-stimulating factor: neuromuscular toxicity is dose-limiting. J Clin Oncol. 1993 Oct;11(10):2010-20. doi: 10.1200/JCO.1993.11.10.2010. PMID 7692001
- [Background] Wiernik PH, Schwartz EL, Strauman JJ, Dutcher JP, Lipton RB, Paietta E. Phase I clinical and pharmacokinetic study of taxol. Cancer Res. 1987 May 1;47(9):2486-93. PMID 2882837
- [Background] Hile ES, Fitzgerald GK, Studenski SA. Persistent mobility disability after neurotoxic chemotherapy. Phys Ther. 2010 Nov;90(11):1649-57. doi: 10.2522/ptj.20090405. Epub 2010 Sep 2. PMID 20813818
- [Background] Jones SE, Erban J, Overmoyer B, Budd GT, Hutchins L, Lower E, Laufman L, Sundaram S, Urba WJ, Pritchard KI, Mennel R, Richards D, Olsen S, Meyers ML, Ravdin PM. Randomized phase III study of docetaxel compared with paclitaxel in metastatic breast cancer. J Clin Oncol. 2005 Aug 20;23(24):5542-51. doi: 10.1200/JCO.2005.02.027. PMID 16110015
- [Background] Dropcho EJ. Neurotoxicity of cancer chemotherapy. Semin Neurol. 2010 Jul;30(3):273-86. doi: 10.1055/s-0030-1255217. Epub 2010 Jun 24. PMID 20577934
- [Background] Dougherty PM, Cata JP, Cordella JV, Burton A, Weng HR. Taxol-induced sensory disturbance is characterized by preferential impairment of myelinated fiber function in cancer patients. Pain. 2004 May;109(1-2):132-42. doi: 10.1016/j.pain.2004.01.021. PMID 15082135
- [Background] Meyer L, Patte-Mensah C, Taleb O, Mensah-Nyagan AG. Neurosteroid 3alpha-androstanediol efficiently counteracts paclitaxel-induced peripheral neuropathy and painful symptoms. PLoS One. 2013 Nov 15;8(11):e80915. doi: 10.1371/journal.pone.0080915. eCollection 2013. PMID 24260511
- [Background] Visovsky C, Collins M, Abbott L, Aschenbrenner J, Hart C. Putting evidence into practice: evidence-based interventions for chemotherapy-induced peripheral neuropathy. Clin J Oncol Nurs. 2007 Dec;11(6):901-13. doi: 10.1188/07.CJON.901-913. PMID 18063548
- [Background] Hershman DL, Lacchetti C, Dworkin RH, Lavoie Smith EM, Bleeker J, Cavaletti G, Chauhan C, Gavin P, Lavino A, Lustberg MB, Paice J, Schneider B, Smith ML, Smith T, Terstriep S, Wagner-Johnston N, Bak K, Loprinzi CL; American Society of Clinical Oncology. Prevention and management of chemotherapy-induced peripheral neuropathy in survivors of adult cancers: American Society of Clinical Oncology clinical practice guideline. J Clin Oncol. 2014 Jun 20;32(18):1941-67. doi: 10.1200/JCO.2013.54.0914. Epub 2014 Apr 14. PMID 24733808
- [Background] Stubblefield MD, Burstein HJ, Burton AW, Custodio CM, Deng GE, Ho M, Junck L, Morris GS, Paice JA, Tummala S, Von Roenn JH. NCCN task force report: management of neuropathy in cancer. J Natl Compr Canc Netw. 2009 Sep;7 Suppl 5:S1-S26; quiz S27-8. doi: 10.6004/jnccn.2009.0078. PMID 19755042
- [Background] Tofthagen C, Visovsky CM, Hopgood R. Chemotherapy-induced peripheral neuropathy: an algorithm to guide nursing management. Clin J Oncol Nurs. 2013 Apr;17(2):138-44. doi: 10.1188/13.CJON.138-144. PMID 23538249
- [Background] Visovsky C, Meyer RR, Roller J, Poppas M. Evaluation and management of peripheral neuropathy in diabetic patients with cancer. Clin J Oncol Nurs. 2008 Apr;12(2):243-7. doi: 10.1188/08.CJON.243-247. PMID 18390460
- [Background] Baron R, Haendler G, Schulte H. Afferent large fiber polyneuropathy predicts the development of postherpetic neuralgia. Pain. 1997 Nov;73(2):231-238. doi: 10.1016/S0304-3959(97)00105-X. PMID 9415510
- [Background] Paice JA. Clinical challenges: chemotherapy-induced peripheral neuropathy. Semin Oncol Nurs. 2009 May;25(2 Suppl 1):S8-19. doi: 10.1016/j.soncn.2009.03.013. PMID 19447319
- [Background] Vadalouca A, Raptis E, Moka E, Zis P, Sykioti P, Siafaka I. Pharmacological treatment of neuropathic cancer pain: a comprehensive review of the current literature. Pain Pract. 2012 Mar;12(3):219-51. doi: 10.1111/j.1533-2500.2011.00485.x. Epub 2011 Jul 29. PMID 21797961
- [Background] Markman M. Chemotherapy-induced peripheral neuropathy: underreported and underappreciated. Curr Pain Headache Rep. 2006 Aug;10(4):275-8. doi: 10.1007/s11916-006-0032-0. PMID 16834942
- [Background] Casanova-Molla J, Grau-Junyent JM, Morales M, Valls-Sole J. On the relationship between nociceptive evoked potentials and intraepidermal nerve fiber density in painful sensory polyneuropathies. Pain. 2011 Feb;152(2):410-418. doi: 10.1016/j.pain.2010.11.012. Epub 2010 Dec 24. PMID 21185650
- [Background] Galer BS. Neuropathic pain of peripheral origin: advances in pharmacologic treatment. Neurology. 1995 Dec;45(12 Suppl 9):S17-25; discussion S35-6. doi: 10.1212/wnl.45.12_suppl_9.s17. PMID 8538882
- [Background] Park SB, Krishnan AV, Lin CS, Goldstein D, Friedlander M, Kiernan MC. Mechanisms underlying chemotherapy-induced neurotoxicity and the potential for neuroprotective strategies. Curr Med Chem. 2008;15(29):3081-94. doi: 10.2174/092986708786848569. PMID 19075655
- [Background] Siao P, Cros DP. Quantitative sensory testing. Phys Med Rehabil Clin N Am. 2003 May;14(2):261-86. doi: 10.1016/s1047-9651(02)00122-5. PMID 12795516
- [Background] Cavaletti G, Frigeni B, Lanzani F, Mattavelli L, Susani E, Alberti P, Cortinovis D, Bidoli P. Chemotherapy-Induced Peripheral Neurotoxicity assessment: a critical revision of the currently available tools. Eur J Cancer. 2010 Feb;46(3):479-94. doi: 10.1016/j.ejca.2009.12.008. Epub 2010 Jan 4. PMID 20045310
- [Background] Xiao WH, Bennett GJ. Chemotherapy-evoked neuropathic pain: Abnormal spontaneous discharge in A-fiber and C-fiber primary afferent neurons and its suppression by acetyl-L-carnitine. Pain. 2008 Apr;135(3):262-270. doi: 10.1016/j.pain.2007.06.001. Epub 2007 Jul 30. PMID 17659836
- [Background] Flatters SJL, Bennett GJ. Studies of peripheral sensory nerves in paclitaxel-induced painful peripheral neuropathy: evidence for mitochondrial dysfunction. Pain. 2006 Jun;122(3):245-257. doi: 10.1016/j.pain.2006.01.037. Epub 2006 Mar 13. PMID 16530964
- [Background] Smith EM. Current methods for the assessment and management of taxane-related neuropathy. Clin J Oncol Nurs. 2013 Feb;17 Suppl:22-34. doi: 10.1188/13.CJON.S1.22-34. PMID 23360700
- [Background] Ocean AJ, Vahdat LT. Chemotherapy-induced peripheral neuropathy: pathogenesis and emerging therapies. Support Care Cancer. 2004 Sep;12(9):619-25. doi: 10.1007/s00520-004-0657-7. PMID 15258838
- [Background] Griffith KA, Dorsey SG, Renn CL, Zhu S, Johantgen ME, Cornblath DR, Argyriou AA, Cavaletti G, Merkies IS, Alberti P, Postma TJ, Rossi E, Frigeni B, Bruna J, Velasco R, Kalofonos HP, Psimaras D, Ricard D, Pace A, Galie E, Briani C, Dalla Torre C, Faber CG, Lalisang RI, Boogerd W, Brandsma D, Koeppen S, Hense J, Storey DJ, Kerrigan S, Schenone A, Fabbri S, Valsecchi MG; CI-PeriNomS Group. Correspondence between neurophysiological and clinical measurements of chemotherapy-induced peripheral neuropathy: secondary analysis of data from the CI-PeriNomS study. J Peripher Nerv Syst. 2014 Jun;19(2):127-35. doi: 10.1111/jns5.12064. PMID 24814100
- [Background] Vas PR, Rayman G. The rate of decline in small fibre function assessed using axon reflex-mediated neurogenic vasodilatation and the importance of age related centile values to improve the detection of clinical neuropathy. PLoS One. 2013 Jul 25;8(7):e69920. doi: 10.1371/journal.pone.0069920. Print 2013. PMID 23936119
- [Background] Krishnan ST, Quattrini C, Jeziorska M, Malik RA, Rayman G. Abnormal LDIflare but normal quantitative sensory testing and dermal nerve fiber density in patients with painful diabetic neuropathy. Diabetes Care. 2009 Mar;32(3):451-5. doi: 10.2337/dc08-1453. Epub 2008 Dec 15. PMID 19074993
- [Background] Vas PR, Rayman G. Validation of the modified LDIFlare technique: a simple and quick method to assess C-fiber function. Muscle Nerve. 2013 Mar;47(3):351-6. doi: 10.1002/mus.23532. Epub 2012 Nov 21. PMID 23169592
- [Background] Krishnan ST, Quattrini C, Jeziorska M, Malik RA, Rayman G. Neurovascular factors in wound healing in the foot skin of type 2 diabetic subjects. Diabetes Care. 2007 Dec;30(12):3058-62. doi: 10.2337/dc07-1421. Epub 2007 Sep 26. PMID 17898089
- [Background] Krishnan ST, Rayman G. The LDIflare: a novel test of C-fiber function demonstrates early neuropathy in type 2 diabetes. Diabetes Care. 2004 Dec;27(12):2930-5. doi: 10.2337/diacare.27.12.2930. PMID 15562209
- [Background] Green AQ, Krishnan S, Finucane FM, Rayman G. Altered C-fiber function as an indicator of early peripheral neuropathy in individuals with impaired glucose tolerance. Diabetes Care. 2010 Jan;33(1):174-6. doi: 10.2337/dc09-0101. PMID 20040675
- [Background] Green AQ, Krishnan ST, Rayman G. C-fiber function assessed by the laser doppler imager flare technique and acetylcholine iontophoresis. Muscle Nerve. 2009 Dec;40(6):985-91. doi: 10.1002/mus.21333. PMID 19768772
- [Background] Kramer HH, Rolke R, Bickel A, Birklein F. Thermal thresholds predict painfulness of diabetic neuropathies. Diabetes Care. 2004 Oct;27(10):2386-91. doi: 10.2337/diacare.27.10.2386. PMID 15451905
- [Background] Wong BJ, Minson CT. Altered thermal hyperaemia in human skin by prior desensitization of neurokinin-1 receptors. Exp Physiol. 2011 Jun;96(6):599-609. doi: 10.1113/expphysiol.2011.057356. Epub 2011 Apr 8. PMID 21478256
- [Background] Minson CT, Berry LT, Joyner MJ. Nitric oxide and neurally mediated regulation of skin blood flow during local heating. J Appl Physiol (1985). 2001 Oct;91(4):1619-26. doi: 10.1152/jappl.2001.91.4.1619. PMID 11568143
- [Background] Persohn E, Canta A, Schoepfer S, Traebert M, Mueller L, Gilardini A, Galbiati S, Nicolini G, Scuteri A, Lanzani F, Giussani G, Cavaletti G. Morphological and morphometric analysis of paclitaxel and docetaxel-induced peripheral neuropathy in rats. Eur J Cancer. 2005 Jul;41(10):1460-6. doi: 10.1016/j.ejca.2005.04.006. PMID 15913989
- [Background] Gilardini A, Avila RL, Oggioni N, Rodriguez-Menendez V, Bossi M, Canta A, Cavaletti G, Kirschner DA. Myelin structure is unaltered in chemotherapy-induced peripheral neuropathy. Neurotoxicology. 2012 Jan;33(1):1-7. doi: 10.1016/j.neuro.2011.10.010. Epub 2011 Nov 4. PMID 22079976
- [Background] Carozzi V, Chiorazzi A, Canta A, Oggioni N, Gilardini A, Rodriguez-Menendez V, Avezza F, Crippa L, Ceresa C, Nicolini G, Bossi M, Cavaletti G. Effect of the chronic combined administration of cisplatin and paclitaxel in a rat model of peripheral neurotoxicity. Eur J Cancer. 2009 Mar;45(4):656-65. doi: 10.1016/j.ejca.2008.10.038. Epub 2008 Dec 16. PMID 19091544
- [Background] Argyriou AA, Koltzenburg M, Polychronopoulos P, Papapetropoulos S, Kalofonos HP. Peripheral nerve damage associated with administration of taxanes in patients with cancer. Crit Rev Oncol Hematol. 2008 Jun;66(3):218-28. doi: 10.1016/j.critrevonc.2008.01.008. Epub 2008 Mar 7. PMID 18329278
- [Background] Authier N, Gillet JP, Fialip J, Eschalier A, Coudore F. Description of a short-term Taxol-induced nociceptive neuropathy in rats. Brain Res. 2000 Dec 29;887(2):239-49. doi: 10.1016/s0006-8993(00)02910-3. PMID 11134612
- [Background] Bennett GJ, Liu GK, Xiao WH, Jin HW, Siau C. Terminal arbor degeneration--a novel lesion produced by the antineoplastic agent paclitaxel. Eur J Neurosci. 2011 May;33(9):1667-76. doi: 10.1111/j.1460-9568.2011.07652.x. Epub 2011 Mar 13. PMID 21395870
- [Background] Boyette-Davis J, Dougherty PM. Protection against oxaliplatin-induced mechanical hyperalgesia and intraepidermal nerve fiber loss by minocycline. Exp Neurol. 2011 Jun;229(2):353-7. doi: 10.1016/j.expneurol.2011.02.019. Epub 2011 Mar 5. PMID 21385581
- [Background] Melli G, Jack C, Lambrinos GL, Ringkamp M, Hoke A. Erythropoietin protects sensory axons against paclitaxel-induced distal degeneration. Neurobiol Dis. 2006 Dec;24(3):525-30. doi: 10.1016/j.nbd.2006.08.014. Epub 2006 Sep 28. PMID 17010629
- [Background] Siau C, Xiao W, Bennett GJ. Paclitaxel- and vincristine-evoked painful peripheral neuropathies: loss of epidermal innervation and activation of Langerhans cells. Exp Neurol. 2006 Oct;201(2):507-14. doi: 10.1016/j.expneurol.2006.05.007. Epub 2006 Jun 22. PMID 16797537
- [Background] Gracias NG, Cummins TR, Kelley MR, Basile DP, Iqbal T, Vasko MR. Vasodilatation in the rat dorsal hindpaw induced by activation of sensory neurons is reduced by paclitaxel. Neurotoxicology. 2011 Jan;32(1):140-9. doi: 10.1016/j.neuro.2010.09.006. Epub 2010 Oct 7. PMID 20932997
- [Background] Pittman SK, Gracias NG, Vasko MR, Fehrenbacher JC. Paclitaxel alters the evoked release of calcitonin gene-related peptide from rat sensory neurons in culture. Exp Neurol. 2014 Mar;253:146-53. doi: 10.1016/j.expneurol.2013.12.011. Epub 2013 Dec 26. PMID 24374060
- [Background] Houghton BL, Meendering JR, Wong BJ, Minson CT. Nitric oxide and noradrenaline contribute to the temperature threshold of the axon reflex response to gradual local heating in human skin. J Physiol. 2006 May 1;572(Pt 3):811-20. doi: 10.1113/jphysiol.2005.104067. PMID 16497714
- [Background] Brain SD, Grant AD. Vascular actions of calcitonin gene-related peptide and adrenomedullin. Physiol Rev. 2004 Jul;84(3):903-34. doi: 10.1152/physrev.00037.2003. PMID 15269340
- [Background] Mahe G, Humeau-Heurtier A, Durand S, Leftheriotis G, Abraham P. Assessment of skin microvascular function and dysfunction with laser speckle contrast imaging. Circ Cardiovasc Imaging. 2012 Jan;5(1):155-63. doi: 10.1161/CIRCIMAGING.111.970418. No abstract available. PMID 22253335
- [Background] Magerl W, Treede RD. Heat-evoked vasodilatation in human hairy skin: axon reflexes due to low-level activity of nociceptive afferents. J Physiol. 1996 Dec 15;497 ( Pt 3)(Pt 3):837-48. doi: 10.1113/jphysiol.1996.sp021814. PMID 9003568
- [Background] Dusch M, Schley M, Rukwied R, Schmelz M. Rapid flare development evoked by current frequency-dependent stimulation analyzed by full-field laser perfusion imaging. Neuroreport. 2007 Jul 16;18(11):1101-5. doi: 10.1097/WNR.0b013e3281e72cff. PMID 17589307
- [Background] Herman RM, Brower JB, Stoddard DG, Casano AR, Targovnik JH, Herman JH, Tearse P. Prevalence of somatic small fiber neuropathy in obesity. Int J Obes (Lond). 2007 Feb;31(2):226-35. doi: 10.1038/sj.ijo.0803418. Epub 2006 Jun 13. PMID 16770330
- [Background] Bickel A, Heyer G, Senger C, Maihofner C, Heuss D, Hilz MJ, Namer B. C-fiber axon reflex flare size correlates with epidermal nerve fiber density in human skin biopsies. J Peripher Nerv Syst. 2009 Dec;14(4):294-9. doi: 10.1111/j.1529-8027.2009.00241.x. PMID 20021571
- [Background] Berghoff M, Kilo S, Hilz MJ, Freeman R. Differential impairment of the sudomotor and nociceptor axon-reflex in diabetic peripheral neuropathy. Muscle Nerve. 2006 Apr;33(4):494-9. doi: 10.1002/mus.20497. PMID 16411196
- [Background] Huang CS, Wang SF, Tsai YF. Axon reflex-related hyperemia induced by short local heating is reproducible. Microvasc Res. 2012 Nov;84(3):351-5. doi: 10.1016/j.mvr.2012.07.003. Epub 2012 Jul 14. PMID 22796314
- [Background] Huang CS, Wang SF, Tsai YF. Increasing acclimation period improves the reproducibility of short-heating local thermal hyperemia. Microvasc Res. 2013 Jan;85:93-8. doi: 10.1016/j.mvr.2012.11.004. Epub 2012 Nov 12. PMID 23154278
- [Background] Nabavi Nouri M, Ahmed A, Bril V, Orszag A, Ng E, Nwe P, Perkins BA. Diabetic neuropathy and axon reflex-mediated neurogenic vasodilatation in type 1 diabetes. PLoS One. 2012;7(4):e34807. doi: 10.1371/journal.pone.0034807. Epub 2012 Apr 17. PMID 22529938
- [Background] Cordovil I, Huguenin G, Rosa G, Bello A, Kohler O, de Moraes R, Tibirica E. Evaluation of systemic microvascular endothelial function using laser speckle contrast imaging. Microvasc Res. 2012 May;83(3):376-9. doi: 10.1016/j.mvr.2012.01.004. Epub 2012 Jan 31. PMID 22326551
- [Background] Tartas M, Bouye P, Koitka A, Durand S, Gallois Y, Saumet JL, Abraham P. Early vasodilator response to anodal current application in human is not impaired by cyclooxygenase-2 blockade. Am J Physiol Heart Circ Physiol. 2005 Apr;288(4):H1668-73. doi: 10.1152/ajpheart.00415.2004. Epub 2004 Nov 24. PMID 15563538
- [Background] Durand S, Fromy B, Bouye P, Saumet JL, Abraham P. Current-induced vasodilation during water iontophoresis (5 min, 0.10 mA) is delayed from current onset and involves aspirin sensitive mechanisms. J Vasc Res. 2002 Jan-Feb;39(1):59-71. doi: 10.1159/000048994. PMID 11844938
- [Background] Dalle-Ave A, Kubli S, Golay S, Delachaux A, Liaudet L, Waeber B, Feihl F. Acetylcholine-induced vasodilation and reactive hyperemia are not affected by acute cyclo-oxygenase inhibition in human skin. Microcirculation. 2004 Jun;11(4):327-36. doi: 10.1080/10739680490449268. PMID 15280072
- [Background] Harris RA, Nishiyama SK, Wray DW, Richardson RS. Ultrasound assessment of flow-mediated dilation. Hypertension. 2010 May;55(5):1075-85. doi: 10.1161/HYPERTENSIONAHA.110.150821. Epub 2010 Mar 29. PMID 20351340
- [Background] de Jongh RT, Clark AD, IJzerman RG, Serne EH, de Vries G, Stehouwer CD. Physiological hyperinsulinaemia increases intramuscular microvascular reactive hyperaemia and vasomotion in healthy volunteers. Diabetologia. 2004 Jun;47(6):978-86. doi: 10.1007/s00125-004-1412-9. Epub 2004 May 28. PMID 15168017
- [Background] Pauling JD, Shipley JA, Raper S, Watson ML, Ward SG, Harris ND, McHugh NJ. Comparison of infrared thermography and laser speckle contrast imaging for the dynamic assessment of digital microvascular function. Microvasc Res. 2012 Mar;83(2):162-7. doi: 10.1016/j.mvr.2011.06.012. Epub 2011 Jul 1. PMID 21763703
- [Background] O'Doherty J, McNamara P, Clancy NT, Enfield JG, Leahy MJ. Comparison of instruments for investigation of microcirculatory blood flow and red blood cell concentration. J Biomed Opt. 2009 May-Jun;14(3):034025. doi: 10.1117/1.3149863. PMID 19566318
- [Background] Rousseau P, Mahe G, Haj-Yassin F, Durand S, Humeau A, Leftheriotis G, Abraham P. Increasing the "region of interest" and "time of interest", both reduce the variability of blood flow measurements using laser speckle contrast imaging. Microvasc Res. 2011 Jul;82(1):88-91. doi: 10.1016/j.mvr.2011.03.009. Epub 2011 Mar 23. PMID 21439303
- [Background] Cracowski JL, Gaillard-Bigot F, Cracowski C, Roustit M, Millet C. Skin microdialysis coupled with laser speckle contrast imaging to assess microvascular reactivity. Microvasc Res. 2011 Nov;82(3):333-8. doi: 10.1016/j.mvr.2011.09.009. Epub 2011 Oct 6. PMID 22001188
- [Background] Blaise S, Roustit M, Millet C, Cracowski JL. Effect of oral sildenafil on skin postocclusive reactive hyperemia in healthy volunteers. Microcirculation. 2011 Aug;18(6):448-51. doi: 10.1111/j.1549-8719.2011.00105.x. PMID 21443694
- [Background] Metzler-Wilson K, Kellie LA, Tomc C, Simpson C, Sammons D, Wilson TE. Differential vasodilatory responses to local heating in facial, glabrous and hairy skin. Clin Physiol Funct Imaging. 2012 Sep;32(5):361-6. doi: 10.1111/j.1475-097X.2012.01137.x. Epub 2012 Apr 12. PMID 22856342
- [Background] Hodges GJ, Traeger JA 3rd, Tang T, Kosiba WA, Zhao K, Johnson JM. Role of sensory nerves in the cutaneous vasoconstrictor response to local cooling in humans. Am J Physiol Heart Circ Physiol. 2007 Jul;293(1):H784-9. doi: 10.1152/ajpheart.00323.2007. Epub 2007 Apr 27. PMID 17468334
- [Background] Vas PR, Green AQ, Rayman G. Small fibre dysfunction, microvascular complications and glycaemic control in type 1 diabetes: a case-control study. Diabetologia. 2012 Mar;55(3):795-800. doi: 10.1007/s00125-011-2417-9. Epub 2011 Dec 23. PMID 22193513
- [Background] Debbabi H, Bonnin P, Ducluzeau PH, Leftheriotis G, Levy BI. Noninvasive assessment of endothelial function in the skin microcirculation. Am J Hypertens. 2010 May;23(5):541-6. doi: 10.1038/ajh.2010.10. Epub 2010 Feb 18. PMID 20168305
- [Background] Tew GA, Klonizakis M, Crank H, Briers JD, Hodges GJ. Comparison of laser speckle contrast imaging with laser Doppler for assessing microvascular function. Microvasc Res. 2011 Nov;82(3):326-32. doi: 10.1016/j.mvr.2011.07.007. Epub 2011 Jul 22. PMID 21803051
- [Background] Wallengren J, Hakanson R. Effects of capsaicin, bradykinin and prostaglandin E2 in the human skin. Br J Dermatol. 1992 Feb;126(2):111-7. doi: 10.1111/j.1365-2133.1992.tb07806.x. PMID 1371395
- [Background] Wong BJ, Fieger SM. Transient receptor potential vanilloid type-1 (TRPV-1) channels contribute to cutaneous thermal hyperaemia in humans. J Physiol. 2010 Nov 1;588(Pt 21):4317-26. doi: 10.1113/jphysiol.2010.195511. PMID 20807792
- [Background] Minson CT, Holowatz LA, Wong BJ, Kenney WL, Wilkins BW. Decreased nitric oxide- and axon reflex-mediated cutaneous vasodilation with age during local heating. J Appl Physiol (1985). 2002 Nov;93(5):1644-9. doi: 10.1152/japplphysiol.00229.2002. PMID 12381749
- [Background] Wiernik PH, Schwartz EL, Einzig A, Strauman JJ, Lipton RB, Dutcher JP. Phase I trial of taxol given as a 24-hour infusion every 21 days: responses observed in metastatic melanoma. J Clin Oncol. 1987 Aug;5(8):1232-9. doi: 10.1200/JCO.1987.5.8.1232. PMID 2887641
- [Background] Takemoto S, Ushijima K, Honda K, Wada H, Terada A, Imaishi H, Kamura T. Precise evaluation of chemotherapy-induced peripheral neuropathy using the visual analogue scale: a quantitative and comparative analysis of neuropathy occurring with paclitaxel-carboplatin and docetaxel-carboplatin therapy. Int J Clin Oncol. 2012 Aug;17(4):367-72. doi: 10.1007/s10147-011-0303-6. Epub 2011 Aug 19. PMID 21850385
- [Background] Tofthagen C, Overcash J, Kip K. Falls in persons with chemotherapy-induced peripheral neuropathy. Support Care Cancer. 2012 Mar;20(3):583-9. doi: 10.1007/s00520-011-1127-7. Epub 2011 Mar 5. PMID 21380613
- [Background] Smith EM, Pang H, Cirrincione C, Fleishman S, Paskett ED, Ahles T, Bressler LR, Fadul CE, Knox C, Le-Lindqwister N, Gilman PB, Shapiro CL; Alliance for Clinical Trials in Oncology. Effect of duloxetine on pain, function, and quality of life among patients with chemotherapy-induced painful peripheral neuropathy: a randomized clinical trial. JAMA. 2013 Apr 3;309(13):1359-67. doi: 10.1001/jama.2013.2813. PMID 23549581
- [Background] Loprinzi CL, Reeves BN, Dakhil SR, Sloan JA, Wolf SL, Burger KN, Kamal A, Le-Lindqwister NA, Soori GS, Jaslowski AJ, Novotny PJ, Lachance DH. Natural history of paclitaxel-associated acute pain syndrome: prospective cohort study NCCTG N08C1. J Clin Oncol. 2011 Apr 10;29(11):1472-8. doi: 10.1200/JCO.2010.33.0308. Epub 2011 Mar 7. PMID 21383290
- [Background] Boyette-Davis JA, Eng C, Wang XS, Cleeland CS, Wendelschafer-Crabb G, Kennedy WR, Simone DA, Zhang H, Dougherty PM. Subclinical peripheral neuropathy is a common finding in colorectal cancer patients prior to chemotherapy. Clin Cancer Res. 2012 Jun 1;18(11):3180-7. doi: 10.1158/1078-0432.CCR-12-0205. Epub 2012 Apr 10. PMID 22496202
- [Background] Donovan D. Management of peripheral neuropathy caused by microtubule inhibitors. Clin J Oncol Nurs. 2009 Dec;13(6):686-94. doi: 10.1188/09.CJON.686-694. PMID 19948466
- [Background] Amara S. Oral glutamine for the prevention of chemotherapy-induced peripheral neuropathy. Ann Pharmacother. 2008 Oct;42(10):1481-5. doi: 10.1345/aph.1L179. Epub 2008 Aug 12. PMID 18698011
- [Background] Argyriou AA, Zolota V, Kyriakopoulou O, Kalofonos HP. Toxic peripheral neuropathy associated with commonly used chemotherapeutic agents. J BUON. 2010 Jul-Sep;15(3):435-46. PMID 20941808
- [Background] Buscemi S, Verga S, Batsis JA, Tranchina MR, Belmonte S, Mattina A, Re A, Rizzo R, Cerasola G. Dose-dependent effects of decaffeinated coffee on endothelial function in healthy subjects. Eur J Clin Nutr. 2009 Oct;63(10):1200-5. doi: 10.1038/ejcn.2009.51. Epub 2009 Jun 24. PMID 19550428
- [Background] Johnson JM, Kellogg DL Jr. Local thermal control of the human cutaneous circulation. J Appl Physiol (1985). 2010 Oct;109(4):1229-38. doi: 10.1152/japplphysiol.00407.2010. Epub 2010 Jun 3. PMID 20522732
- [Background] Cracowski JL, Minson CT, Salvat-Melis M, Halliwill JR. Methodological issues in the assessment of skin microvascular endothelial function in humans. Trends Pharmacol Sci. 2006 Sep;27(9):503-8. doi: 10.1016/j.tips.2006.07.008. Epub 2006 Jul 31. PMID 16876881
- [Background] Smith EM, Cohen JA, Pett MA, Beck SL. The reliability and validity of a modified total neuropathy score-reduced and neuropathic pain severity items when used to measure chemotherapy-induced peripheral neuropathy in patients receiving taxanes and platinums. Cancer Nurs. 2010 May-Jun;33(3):173-83. doi: 10.1097/NCC.0b013e3181c989a3. PMID 20357656
- [Background] Griffith KA, Merkies IS, Hill EE, Cornblath DR. Measures of chemotherapy-induced peripheral neuropathy: a systematic review of psychometric properties. J Peripher Nerv Syst. 2010 Dec;15(4):314-25. doi: 10.1111/j.1529-8027.2010.00292.x. PMID 21199103
- [Background] Smith EM, Beck SL, Cohen J. The total neuropathy score: a tool for measuring chemotherapy-induced peripheral neuropathy. Oncol Nurs Forum. 2008 Jan;35(1):96-102. doi: 10.1188/08.ONF.96-102. PMID 18192158
- [Background] Abraham P, Bourgeau M, Camo M, Humeau-Heurtier A, Durand S, Rousseau P, Mahe G. Effect of skin temperature on skin endothelial function assessment. Microvasc Res. 2013 Jul;88:56-60. doi: 10.1016/j.mvr.2013.04.005. Epub 2013 Apr 27. PMID 23628293
- [Background] Briers JD. Laser Doppler, speckle and related techniques for blood perfusion mapping and imaging. Physiol Meas. 2001 Nov;22(4):R35-66. doi: 10.1088/0967-3334/22/4/201. PMID 11761081
- [Background] Butt KM, Rao TK, Friedman EA, Kountz SL. Venous complications of renal transplantation. Proc Clin Dial Transplant Forum. 1975 Nov;5:77-80. No abstract available. PMID 785466
- [Background] Humeau-Heurtier A, Guerreschi E, Abraham P, Mahe G. Relevance of laser Doppler and laser speckle techniques for assessing vascular function: state of the art and future trends. IEEE Trans Biomed Eng. 2013 Mar;60(3):659-66. doi: 10.1109/TBME.2013.2243449. Epub 2013 Jan 29. PMID 23372072
- [Background] Arora S, Smakowski P, Frykberg RG, Simeone LR, Freeman R, LoGerfo FW, Veves A. Differences in foot and forearm skin microcirculation in diabetic patients with and without neuropathy. Diabetes Care. 1998 Aug;21(8):1339-44. doi: 10.2337/diacare.21.8.1339. PMID 9702444
- [Background] Veves A, Akbari CM, Primavera J, Donaghue VM, Zacharoulis D, Chrzan JS, DeGirolami U, LoGerfo FW, Freeman R. Endothelial dysfunction and the expression of endothelial nitric oxide synthetase in diabetic neuropathy, vascular disease, and foot ulceration. Diabetes. 1998 Mar;47(3):457-63. doi: 10.2337/diabetes.47.3.457. PMID 9519754
- [Background] Krishnan ST, Baker NR, Carrington AL, Rayman G. Comparative roles of microvascular and nerve function in foot ulceration in type 2 diabetes. Diabetes Care. 2004 Jun;27(6):1343-8. doi: 10.2337/diacare.27.6.1343. PMID 15161786
- [Background] Boignard A, Salvat-Melis M, Carpentier PH, Minson CT, Grange L, Duc C, Sarrot-Reynauld F, Cracowski JL. Local hyperemia to heating is impaired in secondary Raynaud's phenomenon. Arthritis Res Ther. 2005;7(5):R1103-12. doi: 10.1186/ar1785. Epub 2005 Jul 19. PMID 16207327
- [Background] Baker N, Green A, Krishnan S, Rayman G. Microvascular and C-fiber function in diabetic charcot neuroarthropathy and diabetic peripheral neuropathy. Diabetes Care. 2007 Dec;30(12):3077-9. doi: 10.2337/dc07-1063. Epub 2007 Sep 5. PMID 17804679
- [Background] Sivaskandarajah GA, Halpern EM, Lovblom LE, Weisman A, Orlov S, Bril V, Perkins BA. Structure-function relationship between corneal nerves and conventional small-fiber tests in type 1 diabetes. Diabetes Care. 2013 Sep;36(9):2748-55. doi: 10.2337/dc12-2075. Epub 2013 Apr 11. PMID 23579181
- [Background] Iredahl F, Lofberg A, Sjoberg F, Farnebo S, Tesselaar E. Non-Invasive Measurement of Skin Microvascular Response during Pharmacological and Physiological Provocations. PLoS One. 2015 Aug 13;10(8):e0133760. doi: 10.1371/journal.pone.0133760. eCollection 2015. PMID 26270037
- [Background] Choi PJ, Brunt VE, Fujii N, Minson CT. New approach to measure cutaneous microvascular function: an improved test of NO-mediated vasodilation by thermal hyperemia. J Appl Physiol (1985). 2014 Aug 1;117(3):277-83. doi: 10.1152/japplphysiol.01397.2013. Epub 2014 Jun 5. PMID 24903917
- [Background] Van Duijnhoven NT, Janssen TW, Green DJ, Minson CT, Hopman MT, Thijssen DH. Effect of functional electrostimulation on impaired skin vasodilator responses to local heating in spinal cord injury. J Appl Physiol (1985). 2009 Apr;106(4):1065-71. doi: 10.1152/japplphysiol.91611.2008. Epub 2009 Feb 19. PMID 19228983
- See also: Gracias N. Paclitaxel alters the function of the small diameter sensory neurons. [Dissertation]. United States--Indiana, Indiana University; 2011. — https://scholarworks.iupui.edu/bitstream/handle/1805/2606/Thesis_Neilia_Gr
- See also: Bruning RS. The mechanisms and functional implications of altered microvascular vasoreactivity in healthy and essential hypertensive men and women [Ph.D.]. Ann Arbor: The Pennsylvania State University; 2013. — http://gradworks.umi.com/35/85/3585564.html